CLINICAL TRIAL: NCT01682798
Title: The Clinical Research on the Efficiency of Yili "Changqing" Pro-ABB Probiotic Yogurt in the Improvement of Human Gastrointestinal Tract System
Brief Title: Study of Yili "Changqing" Pro-ABB Yoghurt in the Improvement of Human Gastrointestinal Tract System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YL/LC-001
Record Dates: First submitted 2012-08-23; First posted 2012-09-11 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Constipation; Dyspepsia; Flatulence; Abdominal Pain
MeSH Terms: conditions — Constipation; Dyspepsia; Flatulence; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Yili "Chang Qing" Pro-ABB yoghurt (Formula 1) (Active Comparator): 100g of Yili "Chang Qing" Pro-ABB yoghurt (Formula 1) will be taken by at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Interventions: Dietary Supplement: Yili "Chang Qing" Pro-ABB yoghurt (Formula 1)
- Placebo yoghurt (Placebo Comparator): 100g of placebo yoghurt (normal yoghurt) will be taken at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Interventions: Dietary Supplement: Placebo yoghurt
- Yili "Chang Qing" Pro-ABB yoghurt (Formula 2) (Active Comparator): 100g of Yili "Chang Qing" Pro-ABB yoghurt (Formula 2) will be taken by at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Interventions: Dietary Supplement: Yili "Chang Qing" Pro-ABB yoghurt (Formula 2)

INTERVENTIONS:
Dietary Supplement: Placebo yoghurt — 100g of placebo yoghurt will be taken at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Arms: Placebo yoghurt
Dietary Supplement: Yili "Chang Qing" Pro-ABB yoghurt (Formula 1) — 100g of Yili "Chang Qing" Pro-ABB yoghurt will be taken by at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Arms: Yili "Chang Qing" Pro-ABB yoghurt (Formula 1)
Dietary Supplement: Yili "Chang Qing" Pro-ABB yoghurt (Formula 2)
  Other Names: 100g of Yili "Chang Qing" Pro-ABB yoghurt will be taken by at 10:00 am and 4:00 pm, respectively; 2 times per day.
  Arms: Yili "Chang Qing" Pro-ABB yoghurt (Formula 2)

SUMMARY:
The purpose of this study is to determine whether Yili "Chang Qing" Pro-ABB yoghurt is effective in improving mild constipation and the intestinal micro-ecology environment & alimentation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 25-45 yrs;
2. Non-specific and/or moderate constipation;
3. Irregular or occasional gastrointestinal disorders (flatulence, gurgling, feeling heavy after eating, abdominal pain);
4. Slow transit or irregular bowels movements (abnormal feces solidity, bowel movements decreased, e.g. every 2-3 days or less than 3 times per week).

Exclusion Criteria:

1. Diagnosed as chronic constipation;
2. Treated gastrointestinal symptoms;
3. Lactose Intolerance;
4. Treatment by analgesic such as aspirin and paracetamol;
5. Had laxatives or other remedies to promote digestion 2 weeks prior to the study start;
6. Consuming dairy products or supplements containing pro/pre-biotic 10 days prior to the study start;
7. Currently suffering from diarrhea.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in constipation condition after 3 weeks | Baseline & 3 weeks

SECONDARY OUTCOMES:
Change in gut resident flora after 3 weeks | Baseline & 3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying An, Ph.D, Study Director — Inner Mongolia Hilo Industrial Group Co., Ltd; Donglian Cai, Principal Investigator — Changhai Hospital of Shanghai, Nutriology Dept.; Xinwang Gao, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Geriatric Medicine Dept..
Locations (2):
- China (2):
  - NanMoFang Community Health Service Center, ChaoYang District, Beijing Municipality
  - JuQuan Community Health Service Center, Gucun, Baoshan District,, Shanghai Municipality